CLINICAL TRIAL: NCT04254536
Title: Changes in Optical Coherence Tomography Leakage Mapping in Diabetic Macular Edema Before and After Treatment With Conbercept
Brief Title: Changes in Optical Coherence Tomography Leakage Mapping in Diabetic Macular Edema After Conbercept Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: OCT-LOR-DME
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Diabetic Macular Edema
Keywords: diebetic macular edema; optical coherence tomography; conbercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Eyes with diabetic macular edema requiring conbercept treatment will be followed up for one month. Before treatment, one week after treatment and one month after treatment, the eyes will be examined by optical coherence tomography (OCT) and optical coherence tomographic angiography (OCTA). The changes of macular edema will be observed and analyzed by OCT leakage mapping software, and the relationship between the changes of macular edema and visual acuity will be analyzed.

DETAILED DESCRIPTION:
1. Research purpose:

   After one month follow-up, we will observe whether OCTleakage mapping can be used as a biomarker to predict the prognosis of DME eyes, and will observe the effect of Conbercept on improving edema and visual acuity of DME eyes.
2. Subjects Number of subjects planned to be recruited: 35

Inclusion criteria:

1. Age ≥ 18
2. Diabetic macular edema eyes treated with conbercept for the first time in 1 week
3. Informed consent of patients and signing of informed consent

Exclusion criteria:

1. High myopia
2. Macular diseases affecting vision
3. Vitreous hemorrhage requiring surgery
4. Patients with anterior segment neovascularization
5. Eye or periocular infection
6. Optic neuropathy and glaucoma
7. Periphlebitis, ophthalmic ischemic syndrome, uveitis, coat's disease, FEVR and other retinal diseases
8. Ametropia and cataract surgery
9. In 3 months, in addition to this treatment of conbercept, other anti VEGF treatment, laser treatment or vitreoretinal surgery were performed
10. Other systemic diseases can not complete follow-up

ELIGIBILITY:
Inclusion Criteria:

1）Age ≥ 18

2) Diabetic macular edema eyes treated with conbercept for the first time in 1 week

3) Informed consent of patients and signing of informed consent

Exclusion Criteria:

1）Myopia ≥ 6.0D

2) Macular diseases affecting vision

3) Vitreous hemorrhage requiring surgery

4) Patients with anterior segment neovascularization

5) Eye or periocular infection

6) Optic neuropathy and glaucoma

7) Periphlebitis, ophthalmic ischemic syndrome, uveitis, coat's disease, FEVR and other retinal diseases

8) Ametropia and cataract surgery

9) In 3 months, in addition to this treatment of conbercept, other anti VEGF treatment, laser treatment or vitreoretinal surgery were performed

10) Other systemic diseases can not complete follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic macular edema in the Renmin Hospital of Wuhan University during the study period
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
central retinal thickness（CRT） | 2020-12
  CRT will be measured by OCT software and the changes before treatment, 1 week after treatment and 1 month after treatment will be compared
best corrected visual acurity(BCVA) | 2020-12
  Compare the changes of BCVA before treatment, 1 week after treatment and 1 month after treatment
low optical ratio(LOR) | 2020-12
  The image will be processed by OCT leakage mapping software, and the changes of LOR will compared before treatment, 1 week after treatment and 1 month after treatment

SECONDARY OUTCOMES:
Ellipsoid Zone | 2020-12
  The continuity of EZ will be judged by OCT image processing, and the changes before treatment, 1 week after treatment and 1 month after treatment will be compared

IPD SHARING:
Plan to Share IPD: Undecided